CLINICAL TRIAL: NCT04108078
Title: Multi-Level Intervention Addressing Intersectional Stigma to Improve HIV Testing in MSM
Brief Title: Promoting Reductions in Intersectional StigMa (PRISM) - GHANA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2000025917; 1R01NR019009-01 (NIH)
Record Dates: First submitted 2019-08-09; First posted 2019-09-27 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: HIV; Stigma
Keywords: HIV; Stigma; Intersectional Stigma; Men who have sex with men
MeSH Terms: conditions — Social Stigma; Homosexuality | interventions — Health Policy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm consists of 1) MSM who receive the intervention (not wait listed) and healthcare facility staff who work at health facilities that have been chosen for the intervention.
  Interventions: Behavioral: Health Policy Plus (HP+); Behavioral: Many Men Many Voices (3MV); Behavioral: HIV Education, Empathy and Empowerment (HIVE3)
- Wait listed (No Intervention): Participants in this arm (MSM and staff at health facilities that were wait listed) will complete assessments, but will receive the intervention after the experimental arm of the study.

INTERVENTIONS:
Behavioral: Health Policy Plus (HP+) — HP+ is a stigma-reduction intervention that is designed to reduce stigmatizing attitudes and beliefs among all workers (clinical and non- clinical) in a healthcare facility.
  Arms: Intervention
Behavioral: Many Men Many Voices (3MV) — 3MV is a group-level HIV prevention intervention designed specifically for use with Black men who have sex with men (MSM). It is a 7- session intervention that is facilitated by trained peers. The intervention has previously been adapted and used with MSM in Ghana.
  Arms: Intervention
Behavioral: HIV Education, Empathy and Empowerment (HIVE3) — The HIVE3 is a telephone-based peer support intervention. It utilizes trained peers, who are also MSM, to provide emotional, informational and affirming support via text message or phone. The intervention was developed specifically for use with MSM in Ghana and demonstrated acceptability and feasibility in a preliminary study in Ghana.
  Arms: Intervention

SUMMARY:
HIV prevalence among men with have sex with men (MSM) in Ghana is at least eight times higher than that of the general population (2%). MSM in Ghana face high levels of stigma due to HIV status (actual or perceived), same-sex behavior, and gender non-conformity. These stigmas are documented barriers to HIV prevention and treatment. In our preliminary work in Ghana (N=137), one-third of MSM had never been tested for HIV. This study is a randomized controlled trial to evaluate the feasibility, acceptability and estimate effect size of a multi-component, multi-level (organizational, interpersonal, and intrapersonal-level) intersectional stigma-reduction intervention to increase HIV testing frequency among MSM in Ghana where HIV, same-sex behavior and gender non-conformity are highly stigmatized. To date, stigma-reduction interventions in Ghana have focused on uni-level targets (e.g., health care facilities (HCFs)) and addressed one type of stigma (e.g., HIV), without engaging the intersectional character of the multiple stigmas that MSM encounter.

Our specific aims are:

1. to evaluate the feasibility and acceptability of a novel multi-component, multi-level intervention to address intersectional stigma.
2. to estimate effect size of the intervention for scale up to a definitive efficacy trial.

Our primary endpoint are:

For MSM: HIV testing, intervention feasibility and acceptability For HCFs: intervention feasibility, acceptability and appropriateness

Our secondary endpoints are:

MSM: Intersectional stigma reduction HCF: Intersectional stigma reduction

This study will combine three theory-based interventions that were previously implemented separately in Ghana for reducing stigma at HCF-level, increasing HIV testing at the peer group-level, and increasing peer social support at the individual-level. Convergence Framework will be used for combining interventions. The ADAPT-ITT framework guides our approach to enhancing the interventions' content on intersectional stigma. To achieve these aims a systematic adaptation that will be used to refine the individually developed HCF, peer- and individual-level interventions to produce a comprehensive multi-level intersectional stigma reduction intervention.

DETAILED DESCRIPTION:
STUDY DESCRIPTION OVERVIEW. Our goal in this study is to determine the feasibility, acceptability and preliminary estimate of effect size of a multi- level intersectional stigma-reduction intervention on HIV testing among MSM in Ghana. This study has two phases: a formative phase and a test phase. The eight-step ADAPT-ITT framework will guide our approach to enhancing the interventions' content to address intersectional stigma and combine the three separate interventions into one multi- level approach. Aim 1 will encompass steps 1-7, leading to the combined multi-level intervention adapted to deepen intersectional stigma content and step 8 in which the study team will conduct a waitlist-controlled RCT of the adapted intervention for feasibility and acceptability. In Aim 2, data generated in the RCT will be used to estimate the effect size of the multi-level intervention on HIV testing among MSM (primary outcome) and intersectional stigma reduction (secondary outcome) among the MSM and HCF staff. In deciding on the RCT with wait-list control was considered with other designs such as factorial designs and a classic RCT design with time and attention-matched controls. It was determined that the RCT with wait-list control was superior to the other designs because our study is premised on the need for combined interventions. Since it is not intended yet to seek to isolate which component of the intervention had the greatest effect on our outcomes, a factorial design was not scientifically justified for our proposed study. Additionally, ethical and budgetary considerations informed our decision to forgo using a structurally equivalent control in favor of a wait-list control for the intervention given the evidence of each interventions' efficacy for reducing stigma among HCF staff and improving HIV testing among MSM.

FORMATIVE PHASE STEP 1: ASSESS Focus group discussions (FGDs) and in-depth interviews (IDIs) will be conducted with MSM and HCF staff to inform the adaptation of the three existing interventions to deepen intersectional stigma content and their integration with each other to address intersectional stigma at multiple levels. FGDs were chosen because of their demonstrated suitability in studies of sexual health and to capitalize on the spontaneous conversational interaction that occurs in groups. This re-creation of the social dynamic with the HCF staff and MSM is critical to the understanding of intersectional stigma from the social organization of these two groups. There are also plans to conduct a limited set of individual interviews to examine more in-depth, topics that elicit intimate personal accounts that may not be suitable for sharing in groups. For example, MSM PLHIV are targeted for IDIs to gain insight into whether and how intersectional stigma experiences influenced their pre- diagnosis prevention behaviors, access to prevention services, timing of HIV testing and linkage to care post-diagnosis.

Qualitatively, the following will be investigated:

1. the drivers and manifestations of HIV, same-sex and gender non-conforming stigmas (intersectional stigma) within HCFs and MSM peer groups
2. how these intersecting stigmas undermine HIV testing
3. perspectives on strategies for reducing intersectional stigma within HCFs and among MSM peer groups. This information will guide to what degree and how these stigmas are addressed within the intervention.

In each study city (Accra and Kumasi), 2-4 FGDs will take place in each with HCF staff and MSM, as well as IDIs with HP+ trainers from the pilot phase (n=10) and MSM with HIV (n=8). The purpose and expectations of involvement in the study will be explained to prospective participants.

STEP 2: DECIDE Guided by the formative research results, the team will meet to discuss what specific intervention activities should be modified to address intersectional stigma. An updated scoping review of research literature to identify innovative evidence-based options to enhance focus on intersecting stigmas, with special attention to technology and social media options. This will include a review of the current intervention activities and discussion of how they can be refined to address intersecting stigmas. In consultation with our civil society partners, the team will then incorporate these changes into the curriculum, identify gaps/errors in logic and make corrections in preparation to conduct a workshop of the intervention with key reference groups.

STEP 3: ADMINISTER After initial modifications, a facilitated simulation workshop of the intervention activities with a combined group of HP+ HCF staff (n=4) and client trainers (n=2) who delivered HP+ in other health facilities in Ghana and MSM (n=8) who received the original 3MV and HIVE3 interventions will take place. Then, the team will conduct a joint workshop session because it is consistent with the concept that the intervention must retain relevance to MSM at all points along the HIV testing pathway, including in the HCF and among their peer-groups. The next step will be produce a revised combined version of the original intervention manuals before the workshop and conduct a series of facilitated simulation exercises with role-play over a 4-day period. Participants will work through each of the intervention levels, focusing on the intersectional stigma content and reviewing our approach to linking the different levels and creating opportunities for safe contact between HCF staff and MSM.

STEP 4: PRODUCE Based on the feedback from the simulation workshop participants and our observations of their engagement with the activities, the study team will determine what content and approaches to incorporate into the adapted intervention manual and which content and processes to edit or forego. In our decision-making process, the study team will give priority consideration to maintaining components that have the highest consistency with scientific literature on intersectional stigma, local cultural relevance, and likelihood to be fun/enjoyable-key requisites for successful intervention uptake.

STEP 5: TOPIC The study team will engage topic experts to review the adapted manual and provide feedback on its congruence with the original intervention and local sociocultural relevance. A copy of the adapted, combined multi-level intervention manual will be provided to the principal investigators of the original separate level interventions. Ghanaian MSM who lead PORSH and YAHR (our two civil-society organization partners that work with Ghanaian MSM) will give feedback that is key to the local cultural relevance and intervention implementation.

STEP 6: INTEGRATE In this step, feedback provided by the topic experts will be taken and summarized in a report that will be distributed to the entire investigative team, including our key local partners. The feedback will be discussed to develop follow-up clarifying questions to the topic experts, as necessary, before making final revisions to the multi-level intervention manual.

STEP 7: TRAIN The study team will also produce a training manual to standardize training and permit future replication of the intervention in other settings. This will provide comprehensive training to study staff whose roles are dedicated to delivering the intervention. In addition, the development of multi-faceted training will take place to facilitate comprehension and retention of training concepts, using strategies that Drs. Nyblade and Nelson has successfully deployed in other HIV prevention research projects. This will include conducting a joint (including teams from both cities) rehearsal of the protocol prior to implementation in the RCT with HCF staff and MSM who are not part of the trial.

RANDOMIZATION PROCEDURES Matched pairing of study facilities: the study will assign four HCFs in each study city to intervention and control groups by matching the size of HCF facility staff censure. In every city, the plan is to first stratify four clinics into a pair of two larger clinics and a pair of two smaller clinics, and then randomly assign one larger and one smaller clinic to either arm. HCFs will be assigned using a randomization sequence created in SAS 9.4 with a 1:1 allocation using random block sizes of four by an independent research assistant. A separate research assistant will open the sealed envelopes to identify group assignment immediately after completion of baseline data collection.

Random assignment of MSM participants. Consented/eligible MSM will be randomized in a 1:1 ratio to intervention versus control arm. A block-randomization approach using a random numbers generator to assign participants to the study arms will be employed, which ensures that the number of participants assigned to the intervention arm in each of the two study cities (or blocks) is approximately equal to the control arm.

ELIGIBILITY:
***RCT***

Inclusion Criteria:

For the RCT, HCF staff are eligible to participate in the study if they are:

* Employed at one of the eight facilities identified for this study and identified with a potential to encounter MSM clients.

For the RCT, MSM are eligible to participate in the study if they are:

* Biologically male at birth
* Currently self-identify as cisgender man
* Report sexual activity with another man at least once within the previous six months and report that they are HIV-negative or status unknown.

Exclusion Criteria:

* HCF staff will be excluded if they anticipate leaving work at the HCF during the study period or have previously participated in HP.
* MSM will be excluded if they plan to move out of the area during the study period.

***Focus Group Discussions (FGDs)***

Inclusion Criteria:

HCF staff are eligible to participate in the FGDs if they are:

* Employed at a study participating facility.

MSM are eligible to participate in FGDs if they are:

* 18 years or older
* Biologically male at birth
* Currently self-identified as cisgender man
* Reported sex with another man at least once within the previous six months. Note: HIV status is not an inclusion criterion for MSM FGD participation.

***In-Depth Interviews (IDI)***

HCF staff are eligible to participate if they are:

* Trained in Health Policy Plus (HP+)
* Have previously delivered HP+ in a Ghanaian HCF

MSM are eligible to participate if:

* 18 years or older
* Biologically male at birth
* Currently self-identified as cisgender man
* Reported sex with another man at least once within the previous six months
* Self-reported that they are living with HIV

Exclusion Criteria:

* Those who do not meet the inclusion criteria listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Part of the study sample will consist only of Ghanaian men who have sex with men. Healthcare facility staff will consist of both men and women. An estimated 70% of healthcare facility staff are female.
Enrollment: 549 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
HIV testing frequency (for MSM) | Change from baseline at 3 months post- intervention
  The intervention will be assessed in the number of completed HIV tests at 3 months compared to baseline. We will combine non-duplicative numbers of self-report and clinic-verified HIV tests (verification is only if an MSM had an HIV test performed at one of the healthcare facilities participating in the multi-level intervention) we are only measuring this outcome with MSM.
HIV testing frequency (for MSM) | Change from baseline at 6 months post- intervention
  The intervention will be assessed in the number of completed HIV tests at 6 months compared to baseline. We will combine non-duplicative numbers of self-report and clinic-verified HIV tests (verification is only if an MSM had an HIV test performed at one of the healthcare facilities participating in the multi-level intervention) we are only measuring this outcome with MSM.

CONTACTS AND LOCATIONS:
Overall Officials: LaRon E. Nelson, PhD, Principal Investigator — Yale School of Nursing
Locations (1):
- University of Ghana School of Public Health, Accra, Greater Accra Region, Ghana

REFERENCES:
- [Derived] Nelson LE, Nyblade L, Torpey K, Logie CH, Qian HZ, Manu A, Gyamerah E, Boakye F, Appiah P, Turner D, Stockton M, Abubakari GM, Vlahov D. Multi-level intersectional stigma reduction intervention to increase HIV testing among men who have sex with men in Ghana: Protocol for a cluster randomized controlled trial. PLoS One. 2021 Nov 29;16(11):e0259324. doi: 10.1371/journal.pone.0259324. eCollection 2021. PMID 34843529